CLINICAL TRIAL: NCT07311265
Title: Effects of a Multi-domain Exercise Program With Motivational Strategies on Anthropometric Variables, Physical Fitness, and Psychological Well-Being of Female Older Adults: A Randomized Controlled Trial
Brief Title: Multi-Domain Exercise Program In Older Women
Acronym: MD-EX Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Oeste de Santa Catarina (Other)
Responsible Party: Principal Investigator, Gracielle Fin, Associate Professor and Researcher in Physical Education and Health Sciences, Universidade do Oeste de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 71244423.0.0000.5367
Record Dates: First submitted 2025-12-08; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy Aging; Overweight and Obesity; Physical Fitness; Psychological Well-being
Keywords: Multidomain exercise; Older women; Physical fitness; Motivation for physical activity; Anthropometric variables; Self-Determination Theory; Randomized controlled trial; Exercise intervention
MeSH Terms: conditions — Overweight; Obesity; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Parallel-group randomized controlled trial with two arms (experimental and control), with participants allocated in a 2:1 ratio and followed for 12 months.
Masking Description: This is an open-label study. Due to the nature of the exercise intervention, neither participants, care providers, investigators, nor outcome assessors were blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Multidomain Exercise Program (Experimental): Participants allocated to the experimental group participated in a supervised 12-month multi-domain exercise program including strength training, aerobic exercises, balance activities, flexibility, and cognitive tasks, combined with motivational and behavioral strategies.
  Interventions: Behavioral: Supervised Multidomain Exercise Program
- Usual Daily Activities (No Structured Exercise) (No Intervention): Participants allocated to the control group maintained their usual daily routines and did not participate in any structured or supervised exercise program during the study period.

INTERVENTIONS:
Behavioral: Supervised Multidomain Exercise Program — Participants engaged in a supervised multi-domain exercise program conducted twice per week for 12 months, with each session lasting approximately 45 minutes. The program included neuromotor activities, muscle-strengthening exercises, aerobic training, balance exercises, flexibility activities, and simple cognitive tasks.
  Exercise intensity was monitored using the Borg Category-Ratio 10 Rating of Perceived Exertion (CR-10), a simple scale that allows participants to rate how hard the exercise feels, along with an affective valence scale to monitor feelings of comfort or discomfort during exercise. Motivational strategies based on Self-Determination Theory (SDT) were incorporated throughout the intervention to support engagement and long-term participation.
  Other Names: Multidomain Training Program
  Arms: Supervised Multidomain Exercise Program

SUMMARY:
The goal of this clinical trial is to learn whether a long-term exercise program can improve physical health and well-being in older women aged 60 years and older who live in the community.

The main questions this study aims to answer are:

* Does taking part in a supervised exercise program lower waist size?
* Does the exercise program improve walking speed, leg strength, and the ability to move safely?
* Does the program improve motivation for physical activity and feelings of support and well-being?

Researchers will compare a Supervised Multi-Domain Exercise Program (intervention group) with Usual Daily Activities (No Structured Exercise) (control group) to see whether the supervised exercise program leads to better physical and psychological outcomes.

Participants will:

* Be randomly assigned to either the exercise program or a control group
* Take part in supervised exercise sessions twice a week for 12 months if assigned to the exercise group
* Complete physical tests, body measurements, and questionnaires about motivation and well-being at the start of the study and after 12 months

DETAILED DESCRIPTION:
This study is a randomized controlled clinical trial designed to examine the effects of a long-term supervised exercise program on physical and psychological outcomes in older women.

A total of 108 women aged 60 years and older who live independently in the community took part in the study. Participants were randomly assigned to one of two groups using a two-to-one ratio. One group was assigned to the Supervised Multi-Domain Exercise Program (intervention group), and the other group was assigned to Usual Daily Activities (No Structured Exercise) (control group).

Participants in the intervention group took part in supervised exercise sessions twice per week for 12 months. Each session lasted about 45 minutes and included a mix of activities focused on strength, walking and movement, balance, flexibility, and simple thinking tasks. Exercise intensity was adjusted to each participant and monitored throughout the program. Motivational strategies were included to support engagement and long-term participation in physical activity.

Participants in the control group continued their usual daily routines and did not take part in any structured or supervised exercise program during the study period.

All participants completed assessments at the start of the study and again after 12 months. These assessments included physical tests, body measurements, and questionnaires related to motivation and well-being. Trained researchers conducted all assessments using standardized procedures.

The study followed established guidelines for clinical trials and was approved by a local Research Ethics Committee. All participants provided written informed consent before taking part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 60 years or older.
* Living independently in the community.
* Ability to walk independently, with or without assistive devices.
* Medical clearance to participate in physical exercise.
* Willingness to participate in the exercise program for 12 months.
* Signed informed consent form.

Exclusion Criteria:

* Presence of severe cardiovascular, respiratory, neurological, or musculoskeletal diseases that contraindicate physical exercise.
* Cognitive impairment that prevents understanding of the study procedures.
* Participation in structured exercise programs more than twice per week in the last three months.
* Recent fractures or surgeries that limit physical activity.
* Any condition that, in the opinion of the research team, could compromise participant safety or adherence to the protocol.

Ages: 60 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who self-identify as women and meet the biological sex eligibility criteria (female at birth) are eligible to participate in this study.
Enrollment: 108 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Waist Girth | Baseline and 12 months
  Change in waist girth after 12 months of intervention, measured in centimeters (cm).
Gait Speed (10-Meter Walk Test) | Baseline and 12 months
  Change in gait speed after 12 months of intervention, assessed using the 10-meter walk test (10MWT), which measures the time needed to walk a distance of 10 meters at a fast and safe pace (seconds).
Lower Limb Functional Strength (Five-Times Sit-to-Stand Test) | Baseline and 12 months
  Change in lower limb functional strength after 12 months of intervention, assessed using the five-times sit-to-stand test (FTSST), which measures the time needed to stand up and sit down five times from a chair (seconds).
Functional Mobility (Timed Up and Go Test) | Baseline and 12 months
  Change in functional mobility after 12 months of intervention, assessed using the Timed Up and Go test (TUG), which measures the time needed to stand up from a chair, walk a short distance, turn around, return, and sit down again (seconds).

SECONDARY OUTCOMES:
Autonomous Regulation for Physical Activity | Baseline and 12 months
  Change in autonomous regulation after 12 months of intervention, assessed using the Treatment Self-Regulation Questionnaire for Physical Activity (TSRQ-PA), a questionnaire that measures reasons for being physically active (score range: 1 to 7).
Controlled Regulation for Physical Activity | Baseline and 12 months
  Change in controlled regulation after 12 months of intervention, assessed using the Treatment Self-Regulation Questionnaire for Physical Activity (TSRQ-PA), which measures externally driven reasons for physical activity (score range: 1 to 7).
Amotivation | Baseline and 12 months
  Change in amotivation after 12 months of intervention, assessed using the Behavioral Regulation in Exercise Questionnaire-3 (BREQ-3), which measures lack of motivation for physical activity (score range: 1 to 5).
Basic Psychological Needs Satisfaction | Baseline and 12 months
  Change in autonomy, competence, and relatedness after 12 months of intervention, assessed using the Basic Need Satisfaction in General Scale (BNSG), which measures satisfaction of basic psychological needs (score range: 1 to 7).
Perceived Health Care Climate | Baseline and 12 months
  Change in perceived autonomy support after 12 months of intervention, assessed using the Health Care Climate Questionnaire (HCCQ), which measures perceived support from health professionals (score range: 1 to 7).

CONTACTS AND LOCATIONS:
Overall Officials: Gracielle Fin, PhD, Principal Investigator — Universidade do Oeste de Santa Catarina
Locations (1):
- Gracielle Fin, Joaçaba, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No